CLINICAL TRIAL: NCT04360330
Title: Phase I Study to Evaluate the Safety and Feasibility of Preoperative Ablative Breast Radiotherapy (SABER) for Selected Early Stage Breast Cancer
Brief Title: SABER Study for Selected Early Stage Breast Cancer
Acronym: SABER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Cristiane Takita, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20190283
Record Dates: First submitted 2020-04-06; First posted 2020-04-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Early-stage Breast Cancer
Keywords: Breast Cancer; Early-stage Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Preoperative SABER (Experimental): * Experimental: Preoperative Stereotactic Ablative Breast Radiotherapy (SABER). Phase I study testing up to 4 dose levels.
  * Non-experimental: Participants will undergo standard partial mastectomy and axillary surgery as per discretion of treating physician 4 to 6 weeks (+ at most 1 week delay) after preoperative SABER is completed.
  Interventions: Radiation: Stereotactic Ablative Breast Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Breast Radiotherapy — Preoperative SABER: Participants will be treated with an assigned dose level of preoperative SABER, delivered in once a day, 5 fractions given on non-consecutive days, over a period of 2 weeks. In this phase I study, starting with dose level II, a dose level of preoperative SABER will be assigned per study dose-escalation design, treating 2 to 6 patients per dose level. The tested doses are the following:
  * Dose Level I: 35 Gy (5 fractions of 7 Gy)
  * Dose Level II (Starting Dose): 40 Gy (5 fractions of 8 Gy)
  * Dose Level III: 45 Gy (5 fractions of 9 Gy)
  * Dose Level IV: 50 Gy (5 fractions of 10 Gy)
  Other Names: SABER

SUMMARY:
The purpose of this study is to find the most effective dose of radiation therapy to give to breast tumors in a shorter period of time, prior to standard partial mastectomy/axillary surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female, ≥ 50 years of age.
2. Oncotype or MammaPrint diagnosis results are required prior to the start of treatment
3. Histologically confirmed invasive breast cancer.
4. Clinical stage T1N0M0.
5. Receptor status: Estrogen-Receptor (ER)/Progesterone-Receptor (PR) positive and Human Epidermal Growth Factor Receptor 2 (HER2) negative.
6. Unifocal breast cancer.
7. Eastern Cooperative Oncology Group (ECOG) 0, 1.
8. Ability to undergo MRI.
9. Women of child-bearing potential (WOCBP) must agree to use adequate contraception or agree to undergo sexual abstinence prior to study entry and for the duration of study participation. WOCBP must have a negative serum or urine pregnancy test at time of enrollment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
10. Ability to understand the investigational nature, potential risks and benefits of the research study and willingness to sign the written informed consent and HIPAA document(s).

Exclusion Criteria:

1. Patients without histologically confirmed invasive breast cancer.
2. Patients without Oncotype or MammaPrint diagnosis results at the start of treatment.
3. Patients with metastatic disease.
4. ECOG 2, 3, 4.
5. Patients that are unable to undergo MRI.
6. Prior history of radiation to the chest.
7. History of collagenous disease (systemic lupus erythematosus, scleroderma, dermatomyositis).
8. Any serious medical or psychiatric illness/condition likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment.
9. Diagnosis of another primary malignancy within the last 5 years with the exception of non-melanoma skin cancer.
10. Patients unable to consent, who are pregnant or nursing, or are prisoners.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-08-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) of Pre-Operative SABER | Up to 13 Weeks
  The recommended phase 2 dose (RP2D) of pre-operative SABER therapy will be established as the highest dose level tested for which no more than 1 out of 6 patients experience dose-limiting toxicity (DLT). Adverse Events (AEs) including DLTs will be evaluated by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Number of Participants Experiencing Treatment-Related Toxicity | Up to 13 weeks
  Number of participants experiencing treatment-related toxicity by type and grade including adverse event (AEs), serious adverse events (SAEs) and dose-limiting toxicities (DLTs). Toxicity will be evaluated using the NCI CTCAE version 5.0.
Percentage of participants with Complete Pathological Response (pCR) | Up to 9 weeks
  pCR will be defined as a negative pathologic specimen for invasive carcinoma. The specimen used for evaluation will be the tissue samples obtained from standard of care partial mastectomy and axillary surgery as per discretion of treating physician.
Cosmesis Evaluation | 1, 6 ,12 and 24 months post-therapy, up to 2.5 years
  Participant cosmesis will be evaluated-by-physician at 1, 6,12 and 24 months post-SABER therapy and post-surgical follow-up, using the Harvard 4-point ordinal scale (excellent, good, fair, and poor).
Participant-Reported Health-Related Quality of Life (HR-QoL) | 1, 6 ,12 and 24 months post-therapy, up to 2.5 years
  The Breast Cancer Treatment Outcome Scale (BCTOS) questionnaire will be used to assess participant-reported health-related quality of life (HR-QoL) at 1, 6 12, 24 months post-SABER therapy and post-surgical follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Takita, MD, MBA, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No